CLINICAL TRIAL: NCT00051571
Title: A Phase II Study Using SGN-15 (cBR96-Doxorubicin Immunoconjugate) in Combination With Docetaxel for the Treatment of Advanced Stage or Recurrent Non-Small Cell Lung Carcinoma
Brief Title: Safety/Efficacy Study of Immunoconjugate With Docetaxel in Non-small Cell Lung Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SG0002-015; NCT00031603 (obsolete NCT alias)
Record Dates: First submitted 2003-01-13; First posted 2003-01-15 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

INTERVENTIONS:
Drug: SGN-15
Drug: Docetaxel

SUMMARY:
This randomized phase II clinical trial evaluates the combination of a monoclonal antibody-based drug (SGN-15) with a chemotherapeutic agent compared to chemotherapy given alone in patients with non-small cell lung cancer that has failed at least one prior systemic therapy. The objective of the study is to determine the safety and clinical benefit, as measured by tumor response and quality of life, to the combination regimen.

Monoclonal antibody therapy has been used in other types of cancer to target therapy to the tumor, thereby allowing for the chemotherapeutic agent to have a lesser effect on normal, healthy tissue.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with pathologically confirmed NSCLC which is metastatic or recurrent (non-resectable), who have failed at least one but no more than two prior therapies for advanced stage disease or have a recurrence within 6 months of completing adjuvant chemotherapy.

Lewis-y antigen expression documented by immunohistochemistry for all patients.

Patients must have:

* Bidimensionally or unidimensionally measurable disease on the basis of physical exam or imaging studies, or
* Evaluable disease: bone metastases defined on bone scan or malignant pleural effusion

Performance status ≤ 2 (ECOG scale) with a life expectancy of at least 3 months

Patients must be at least four weeks from prior treatment (chemotherapy, hormonal therapy, or definitive radiotherapy)

EXCLUSION CRITERIA:

Prior therapy with TAXOTERE (docetaxel)

Cumulative anthracycline exposure > 300 mg/m2.

More than one primary malignancy with the exception of:

* Non-melanoma skin cancer
* In situ carcinoma of the cervix
* Localized prostate cancer
* Completely resected stage I or II disease with no evidence of recurrent cancer from which the patient has remained disease free for more than 3 years.

Uncontrolled significant non-malignant disease (e.g. congestive heart failure, bleeding, renal failure, hepatic failure).

Uncontrolled, symptomatic brain metastasis.

Peripheral neuropathy > grade 2.

Concomitant therapy with other anti-neoplastic agents or experimental agents except for small volume radiation to a solitary bony metastasis.

Active viral, bacterial or systemic fungal infections including known HIV or Hepatitis B or C.

Women who are pregnant or breastfeeding

Any serious underlying medical condition, which would impair the ability of the patient to receive the planned treatment including prior allergic reactions to recombinant human or murine proteins.

Dementia or altered mental status that would prohibit the understanding and rendering of informed consent.

Patients with uncontrolled peptic ulcer disease will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sandler, MD, Study Director — Seagen Inc.
Locations (9):
- United States (9):
  - UCLA Medical Center, Los Angeles, California
  - Bendheim Cancer Center, Greenwich, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - University of Chicago, Chicago, Illinois
  - Providence Health System, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Virginia Mason Research Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington